CLINICAL TRIAL: NCT05760313
Title: A Phase 2 Dose Finding Study Evaluating the Safety and Efficacy of Linaclotide in Pediatric Subjects 6 Months to Less Than 2 Years of Age With Functional Constipation (FC).
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity in Pediatric Participants (Age 6 Months to <2 Years) With Functional Constipation Who Are Treated With Linaclotide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-862; 2022-501947-34-00 (Other: EU CT)
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Functional Constipation
Keywords: Linaclotide; pediatric functional constipation; Linzess
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1, Linaclotide Dose A (Experimental): Linaclotide Dose A capsules, mixed with water and administered orally, once daily for 4 weeks
  Interventions: Drug: Linaclotide
- Part 1, Linaclotide Dose B (Experimental): Linaclotide Dose B capsules, mixed with water and administered orally, once daily for 4 weeks
  Interventions: Drug: Linaclotide
- Part 1, Linaclotide Dose C (Experimental): Linaclotide Dose C capsules, mixed with water and administered orally, once daily for 4 weeks
  Interventions: Drug: Linaclotide
- Part 2, Linaclotide (Experimental): Participants will receive Linaclotide capsules mixed with water and administered orally in Part 2 for 4 weeks.
  Interventions: Drug: Linaclotide
- Part 2, Placebo (Experimental): Participants will receive placebo capsules mixed with water and administered orally in Part 2 for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide — Capsule; oral
  Other Names: Linzess
  Arms: Part 1, Linaclotide Dose A; Part 1, Linaclotide Dose B; Part 1, Linaclotide Dose C; Part 2, Linaclotide
Drug: Placebo — Capsule; oral
  Arms: Part 2, Placebo

SUMMARY:
Functional constipation (FC) is a common healthcare problem in children of all ages, potentially due to genetic predisposition, inadequate fiber and fluid intake, and immobility. Currently, there are no pharmacological therapies approved for the treatment of FC. This study will assess adverse events and change in disease activity with linaclotide therapy in participants with FC.

Linaclotide is an approved drug being developed for the treatment of FC in pediatric patients who meet modified Rome IV criteria for childhood FC. In Part 1 of this study, participants are placed in 3 groups, which occur consecutively. Each group receives a different dosage of linaclotide. In Part 2 of the study, participants will be randomly assigned to receive either linaclotide or placebo. There is a 1 in 2 chance that participants will be assigned to placebo. Up to 30 and at least 18 pediatric participants 6 months to less than 2 years of age with FC will be enrolled in the study at approximately 38 sites worldwide.

Participants will receive oral solution of linaclotide prepared from capsule by parent/guardian once daily for 4 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be 6 months to less than 1 year and 11 months old, at the time the legally authorized representative (LAR)/parent/guardian signs the informed consent in alignment with local requirements.
* The LAR/parent/guardian who will be completing the electronic diary (eDiary) is able to read and understand the assessments in the eDiary device and must undergo training.
* Participant meets Rome IV criteria for functional constipation (FC): for at least 1 month before Screening (Visit 1), the participant must meet 2 or more of the following:

  * 2 or fewer defecations per week (with each defecation occurring in the absence of any laxative, suppository, or enema use during the preceding 24 hours)
  * History of excessive stool retention
  * History of painful or hard bowel movements (BMs)
  * History of large-diameter stools
  * Presence of a large fecal mass in the rectum
* LAR/Parent/Guardian is willing to discontinue any laxatives used before the Preintervention Visit in favor of the protocol-permitted rescue medicine.

Exclusion Criteria:

* Participant has conditions that could interfere with drug absorption, including, but not limited to, short bowel syndrome.
* History of clinically significant medical conditions or any other reason that the investigator determines would interfere with the individual's participation in this study or would make the participant an unsuitable candidate to receive study drug.
* Participant has history of:

  * Celiac disease, or positive serological test for celiac disease or the condition is suspected but has not been ruled out by endoscopic biopsy
  * Cystic fibrosis
  * Hypothyroidism that is untreated or treated with thyroid hormone at a dose that has not been stable for at least 3 months prior to Screening (Visit 1)
  * Down's syndrome or any other chromosomal disorder
  * Active anal fissure (investigator has confirmed an active anal fissure and participant reports known anal fissure symptoms [i.e., streaks of blood on the stool or on diaper or toilet paper and pain/crying with bowel movement within 2 weeks prior to Screening]). (Note: Anal fissures that have resolved at least 2 weeks prior to screening would not be exclusionary). However, if in the investigator's opinion, an anal fissure(s) may be the primary cause of participant's Rome IV FC criteria, the subject would not be eligible to participate in the study.
  * Anatomic malformations (e.g., imperforate anus, anal stenosis, anterior displaced anus)
  * Intestinal nerve or muscle disorders (e.g., Hirschprung disease, visceral myopathies, visceral neuropathies)
  * Neuropathic conditions (e.g., spinal cord abnormalities, neurofibromatosis, tethered cord, spinal cord trauma)
  * Lead toxicity, hypercalcemia
  * Inflammatory bowel disease
  * Lactose intolerance that is associated with symptoms which could confound the assessments in this study
  * History of cancer. (Note: Participants with a history of cancer are allowed provided that the malignancy has been in a complete remission before enrollment/randomization (Visit 3). A complete remission is defined as the disappearance of all signs of cancer in response to treatment)

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (38):
- United States (18):
  - Velocity Clinical Research - Phoenix /ID# 263871, Phoenix, Arizona
  - HealthStar Research of Hot Springs PLLC /ID# 251553, Hot Springs, Arkansas
  - Advanced Research Center /ID# 248763, Anaheim, California
  - Kindred Medical Institute - Corona /ID# 251535, Corona, California
  - Velocity Clinical Research Washington DC /ID# 263872, Washington D.C., District of Columbia
  - Prohealth Research Center /ID# 248696, Doral, Florida
  - South Miami Medical & Research Group Inc. /ID# 248765, Miami, Florida
  - Valencia Medical & Research Center /ID# 251533, Miami, Florida
  - Velocity Clinical Research Macon /ID# 263959, Macon, Georgia
  - Velocity Clinical Research - Lafayette /ID# 263873, Lafayette, Louisiana
  - Frederick County Pediatrics /ID# 251555, New Market, Maryland
  - Michigan Center of Medical Research /ID# 253536, Farmington Hills, Michigan
  - Velocity Clinical Research- Hastings Nebraska /ID# 260932, Hastings, Nebraska
  - Coastal Pediatric Research - West Ashley B /ID# 248693, Charleston, South Carolina
  - Coastal Pediatric Research - Summerville /ID# 253534, Summerville, South Carolina
  - Houston Clinical Research Associates /ID# 261571, Houston, Texas
  - Prime Clinical Research - Mansfield - East Broad Street /ID# 262947, Mansfield, Texas
  - ClinPoint Trials /ID# 251534, Waxahachie, Texas
- Bulgaria (5):
  - UMHAT Sveti Georgi /ID# 250808, Plovdiv
  - UMHAT Kanev /ID# 248931, Rousse
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 251232, Sofia
  - Specialized Hospital For Active Treatment Of Children Diseases Prof. Ivan Mitev /ID# 251229, Sofia
  - Nova Clinic /ID# 249023, Varna
- Croatia (4):
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 252798, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 252796, Zagreb, City of Zagreb
  - Klinika za dječje bolesti Zagreb /ID# 252792, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 252795, Osijek, County of Osijek-Baranja
- Germany (3):
  - Universitaetsklinikum Muenster /ID# 251965, Münster, North Rhine-Westphalia
  - Kinderarztpraxis Dr. Froehlich /ID# 252050, Forchheim
  - HELIOS Klinikum Wuppertal /ID# 249022, Wuppertal
- Debreceni Egyetem-Klinikai Kozpont /ID# 250793, Debrecen, Hajdú-Bihar, Hungary
- Serbia (3):
  - Institut za zdravstvenu zastitu majke i deteta Srbije Dr Vukan Cupic /ID# 252485, Belgrade, Beograd
  - University Children's Hospital 'Tirsova' /ID# 252483, Belgrade, Beograd
  - Institute for Child and Youth Health Care of Vojvodina /ID# 252482, Novi Sad
- United Kingdom (4):
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 252298, London, Greater London
  - Great Ormond Street Children's Hospital /ID# 253333, London, Greater London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 252299, Norwich, Norfolk
  - Russells Hall Hospital /ID# 252660, Dudley

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://www.abbvieclinicaltrials.com/study/?id=M21-862

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Linaclotide 9 µg (Part 1): Linaclotide capsules, mixed with water (or apple juice or apple sauce) and administered orally, once daily for 4 weeks in Part 1.
  Linaclotide: Capsule; oral
- Double-Blind Placebo (Part 2): Participants will receive placebo capsules mixed with water (or apple juice or apple sauce) and administered orally in Part 2 for 4 weeks.
  Placebo: Capsule; oral
- Double-Blind Linaclotide 9 µg (Part 2): Participants will receive Linaclotide capsules mixed with water (or apple juice or apple sauce) and administered orally in Part 2 for 4 weeks.
  Linaclotide: Capsule; oral
Period: Overall Study
Arm/Group | Open-Label Linaclotide 9 µg (Part 1) | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2)
Started | 7 | 6 | 6
Completed | 6 | 6 | 5
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population was used for all efficacy and baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-Label Linaclotide 9 µg (Part 1) | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2) | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: months] | 17.1 (5.49) | 15.8 (5.34) | 18.5 (4.97) | 17.1 (5.27)
Age, Customized [Count of Participants; unit: Participants]
  6 - <12 months | 1 | 1 | 1 | 3
  12 - 24 months | 6 | 5 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 1 | 8
  Male | 2 | 4 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 2 | 11
  Not Hispanic or Latino | 3 | 1 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 4 | 6
  White | 6 | 4 | 2 | 12
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Spontaneous Bowel Movement (SBM) Frequency Rate (SBMs/Week) During the Study Intervention Period
Description: An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the BM or the calendar day before the BM. The caregiver/parent/guardian/legally authorized representative (LAR) will complete the electronic diary (eDiary), providing data for the SBM frequency rate up to the last dose date equivalent to the 4-week SBM frequency rate.
Time Frame: Baseline to Week 4
Population: The ITT population was used for all efficacy and baseline analyses.
Measure: Mean (Standard Deviation); unit: SBMs/Week
Arm/Group | Open-Label Linaclotide 9 µg (Part 1) | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2)
Number analyzed (Participants) | 7 | 6 | 6
SBMs/Week
  Observed by the LAR/Parent/Guardian/Caregiver | 3.181 (0.9563) | 2.503 (1.3791) | 0.246 (0.7035)
  All Reported by the LAR/Parent/Guardian/Caregiver | 3.371 (0.9858) | 2.577 (1.4293) | 0.895 (1.1475)

2. Primary Outcome: Change From Baseline in Stool Consistency (Bristol Stool Form Scale) During the Study Intervention Period
Description: The caregiver/parent/guardian/legally authorized representative (LAR) will rate and record in an eDiary the consistency of the stool for each BM using the Bristol Stool Form 7-point scale in which 1=Separate hard lumps, like nuts (hard to pass); 2=Sausage-shaped, but lumpy; 3=Like a sausage but with cracks on its surface; 4=Like a sausage or snake, smooth and soft; 5=Soft blobs with clear cut edges (easy to pass); 6=Fluffy pieces with ragged edges, a mushy stool; and 7=Watery, no solid pieces, entirely liquid.
Time Frame: Baseline to Week 4
Population: The ITT population was used for all efficacy and baseline analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Linaclotide 9 µg (Part 1) | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2)
Number analyzed (Participants) | 7 | 6 | 6
units on a scale | 0.845 (2.1137) | 1.062 (0.8043) | 1.201 (1.0192)

3. Primary Outcome: Change From Baseline in Straining During the Study Intervention Period
Description: Straining for each LAR/parent/guardian/caregiver-observed BM the child passes was collected daily in the eDiary device, using a 4-point scale (0 = No, not at all; 1 = Yes, a little; 2 = Yes, a lot; 3 = I don't know) based on two questions (did he/she grunt or make a face like he/she was straining). Lower value represents a better outcome and "I don't know" is considered as a missing response. The subject's average straining score for each caregiver-observed BM was derived based on the average of non-missing responses of the two straining questions. The participant's straining score in the 4-week Study Intervention Period was the average of the non-missing average straining scores from all caregiver-observed SBMs during the 4-week Study Intervention Period. If a subject had no caregiver-observed SBMs at baseline, then the baseline straining score reported by the caregiver was missing and, therefore, that subject was not included in the change from baseline straining analysis.
Time Frame: Baseline to Week 4
Population: The ITT population was used for all efficacy and baseline analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Linaclotide 9 µg (Part 1) | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2)
Number analyzed (Participants) | 7 | 6 | 6
score on a scale | -1.087 (0.6511) | -0.821 (0.9659) | -0.561 (0.3779)

4. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Time Frame: Up to Week 5
Population: The SA analysis population was used for safety analyses.
Measure: Number; unit: participants
Arm/Group | Open-Label Linaclotide 9 µg (Part 1) | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2)
Number analyzed (Participants) | 7 | 6 | 6
participants | 3 | 1 | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 72.5, 76.5, and 77 days for Double-Blind Placebo, Double-Blind Linaclotide 9 µg (Part 2), and Open-Label Linaclotide 9 µg (Part 1), respectively.
Groups:
- Double-Blind Placebo (Part 2): Participants will receive placebo capsules mixed with water (or apple juice/apple sauce) and administered orally in Part 2 for 4 weeks.
  Placebo: Capsule; oral
- Double-Blind Linaclotide 9 µg (Part 2): Participants will receive Linaclotide capsules mixed with water (or apple juice/apple sauce) and administered orally in Part 2 for 4 weeks.
  Linaclotide: Capsule; oral
- Open-Label Linaclotide 9 µg (Part 1): Linaclotide capsules, mixed with water (or apple juice/apple sauce) and administered orally, once daily for 4 weeks in Part 1.
  Linaclotide: Capsule; oral
Arm/Group | Double-Blind Placebo (Part 2) | Double-Blind Linaclotide 9 µg (Part 2) | Open-Label Linaclotide 9 µg (Part 1)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Placebo (Part 2) (N=6) | Double-Blind Linaclotide 9 µg (Part 2) (N=6) | Open-Label Linaclotide 9 µg (Part 1) (N=7)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTITIS MEDIA ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT05760313/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT05760313/SAP_001.pdf